CLINICAL TRIAL: NCT05629884
Title: Efficacy of a Physical and Respiratory Rehabilitation Program (COPERIA-REHAB) for Patients With Persistent COVID-19 (SARS-CoV-2).
Brief Title: Efficacy of a Physical and Respiratory Rehabilitation Program for Patients With Persistent COVID-19 (SARS-CoV-2).
Acronym: COPERIA-REHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: University of Vigo (Other); Galician South Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COPERIA-REHAB
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19 Recurrent; Cognitive Dysfunction; Fatigue
Keywords: COVID-19; SARS-CoV-2; Persistent Covid; Cardiac rehabilitation; Respiratory rehabilitation; Physical rehabilitation
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): This group will perform the rehabilitation from home or from the gym following online instructions in the COPERIA platform.
  Interventions: Other: COPERIA-REHAB
- Control arm (No Intervention): This control arm will train at the rehabilitation service or at home following the instructions provided by the rehabilitation service.

INTERVENTIONS:
Other: COPERIA-REHAB — After the randomization of the patient there will be some preliminary sessions where the means of self-monitoring training and the Borg 1/10 effort scale will be explained and training videos will be shown. Doubts will also be answered.
  Afterwards, training will start through the COPERIA-REHAB platform, which will last 8 weeks (6 days per week).
  Arms: Experimental arm

SUMMARY:
The pandemic caused by SARS-CoV-2 infection has resulted, in addition to the well-known acute symptoms, in the emergence of a plethora of persistent, diffuse and heterogeneous symptoms such as fatigue, shortness of breath and cognitive dysfunction among others, that have come to be called persistent COVID. Patients have reported that physical activity, stress and sleep disturbances often trigger exacerbations of their symptoms related by some authors to the so-called Post Exertional Malaise (PEM) characteristic of Myalgic Encephalomyelitis. Similarly, by analogy with other pathologies, it has been hypothesized that optimal exercise prescription would benefit these people with persistent COVID-19 symptoms but in practice, the rehabilitation of these patients runs the risk of collapsing respiratory and physical rehabilitation services.

This is why COPERIA proposes the construction of a platform for respiratory, cardiac and muscular telerehabilitation, to compare with face-to-face rehabilitation treatment and to try to predict the influence of physical activity in the prediction of PEM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years of age.
* Patients with a diagnosis according to WHO criteria of persistent COVID-19 until 03/28/2022
* Patients with a Post Covid Functional Status (PCFS) ≥ 2.
* Patients who present a need for physical rehabilitation and agree to perform it.
* Patients with capacity to consent and who agree to participate in the study.
* Patients who know how to use Smartphone and/or Tablet and have at least one of these devices.
* Patients who have access to the rehabilitation tools at home or are willing to go to the gyms proposed in the study to perform the rehabilitation exercises.

Exclusion Criteria:

* Minors or persons judicially incapacitated.
* Previous neurological or psychiatric pathology involving neuropsychological compromise.
* Active Covid19 infection.
* Home oxygen therapy > 16 hours or home Cpap- Bipap.
* Previous diagnosis of arrhythmia or blockage.
* Previous coronary pathology.
* Decompensated renal or metabolic disease.
* Signs or symptoms of unknown cardiac disease.
* Undergoing another physical or cognitive rehabilitation process at the time of inclusion.
* Patients who do not agree to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-12-14 (Estimated); Primary Completion 2023-11-14 (Estimated); Study Completion 2023-11-14 (Estimated)

PRIMARY OUTCOMES:
Six Minutes Walking test | 8 weeks
  The 6-min walk test is a standard in cardiac rehabilitation, serving both to ecologically determine the patient's functional status and to make recommendations regarding the intensity of rehabilitative exercise. The patient is asked to run the maximum distance he/she can in 6 minutes. The length of one of the hospital corridors has been previously measured so that by counting the number of times the patient walks the distance covered is determined. In addition to the number of meters, the heart rate is monitored by means of a pectoral band, and the saturation level by means of a pulse oximeter; the BP is evaluated before and after the test. In the context of functional assessment of Persistent COVID, it has been used for the evaluation of the impact of rehabilitation measures.

SECONDARY OUTCOMES:
mMRC dyspnea scale | 8 weeks
  The MRC shortness of breath scale consists of five statements that describe almost the entire range of respiratory disability, from none (Grade 1) to almost complete disability (Grade 5). It can be self-administered by asking subjects to choose the statement that best describes their condition, e.g., "'I am only short of breath with strenuous exertion" (Grade 1) or "I am so short of breath that I cannot leave the house" (Grade 5). Alternatively, it can be administered by an interviewer asking the questions, such as "Are you short of breath when rushing on level ground or when climbing a gentle slope?" (Grade 2). The score is the number that best matches the patient's activity level.
SF-36 Health Questionnaire | 8 weeks
  The SF-36 Health Questionnaire is composed of 36 items that assess both positive and negative states of health. The 36 items of the instrument cover the following scales: Physical Function, Physical Role, Bodily Pain, General Health, Vitality, Social Function, Emotional Role, and Mental Health. Additionally, the SF-36 includes a transition item that asks about the change in general health status from the previous year.
Maximal Handgrip Strenght | 8 weeks
  Handgrip strength (HGS) is measured by a handgrip dynamometer and is considered an indicator of overall muscle strength. Low muscle strength, also known as dynapenia is an important indicator of health status, as well as an indicator of sarcopenia. Maximal grip strength is determined by performing three grip attempts at maximum power.
1 Minute Sit to Stand test | 8 weeks
  Consists of sitting down and getting up from a chair without resting the hands as many times as possible for 1 minute with the patient connected to the saturator and monitored with a chest strap. The minute is timed, the number of repetitions performed is counted, the oxygen saturation value and heart rate are observed and the patient waits 1 minute after the exercise to record again the recovery of the basal parameters.
P maximal inspiratory and P maximal expiratory | 8 weeks
  These tests will be performed by the Pneumology Service. The measurement of maximal inspiratory and expiratory pressures are well tolerated and relatively easy to perform, they allow estimating the neuromuscular function of the diaphragm, as well as the abdominal, intercostal and accessory muscles. In general terms, the Pimax test estimates the strength of inspiratory muscles (diaphragm) and the Pemax test estimates the strength of abdominal and intercostal muscles. The tests consist of the patient having to generate maximum inspiratory and expiratory pressures against an occluded mouthpiece.
Insomnia Severity Index. | 8 weeks
  This instrument for the assessment of insomnia consists of 7 questions that are rated between 0 and 4 points. It evaluates both the insomnia of conciliation, maintenance and early awakening, as well as its functional repercussions during the day.

OTHER OUTCOMES:
Age | 8 weeks
  Years
Sex | 8 weeks
  Male, Female
Body mass index | 8 weeks
  kg/m^2
Current treatment | 8 weeks
  Treatment taken by the patient at the time of the study.
Date of PCR + SARS-CoV-2 | 8 weeks
  DD-MMM-YYYY
Epidemic wave | 8 weeks
  Of the 7 waves of COVID-19 that have occurred in Spain, a description will be given of the wave to which the infection of each patient included belonged. First, second, third, fourth, fifth, sixth, seventh, eighth, ninth or tenth wave.
Vaccination status at the time of infection | 8 weeks
  Number of vaccine doses at the time of infection
FVC | 8 weeks
  Is the maximum volume of air exhaled, with the maximum possible effort, starting from a maximum inspiration in ml.
FEV1 | 8 weeks
  The volume of air expelled during the first second of forced expiration in ml
FEV1/FVC | 8 weeks
  Expressed as a percentage (%), it indicates the proportion of the FVC that is expelled during the first second of the forced expiratory maneuver.
CO diffusion test | 8 weeks
  To evaluate the transfer of oxygen from the alveolar space to the hemoglobin of the erythrocytes contained in the pulmonary capillaries. Effective alveolar-capillary area available for gas transfer in the lung. (%)

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Galicia Sur Health Research Institute (IISGS) - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - School of Telecommunication Engineering (University of Vigo), Vigo, Pontevedra
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - S.S. Computer Engineering (University of Vigo), Ourense